CLINICAL TRIAL: NCT05304702
Title: Lung Injury (Pulmonary Edema) in COVID-19: Treatment With Furosemide and Negative Fluid Balance (NEGBAL): a Case-Control Study
Brief Title: Lung Injury (Pulmonary Edema) in COVID-19: Treatment With Furosemide and Negative Fluid Balance (NEGBAL)
Status: Completed | Type: Observational
Sponsor: Clinica Colon (Other)
Responsible Party: Principal Investigator, José Luis Francisco Santos, Chief of Intensive Care Unit, Clinica Colon
Other Study IDs: UTI-ESI-002
Record Dates: First submitted 2022-03-17; First posted 2022-03-31 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
Keywords: furosemide; edema; volume overload; diuretic; NEGBAL - Negative Fluid Balance; COVID-19
MeSH Terms: conditions — COVID-19; Edema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NEGBAL: Negative Fluid Balance (NEGBAL) Approach:
  COVID-19 patients with tomographic detection of pulmonary edema (dilated superior vena cava, large pulmonary arteries, diffuse interstitial infiltrates with Kerley lines, and dilated right ventricle or dilated cardiac axis) treated with NEGBAL approach. This consisted of oral hydric restriction and use of diuretics (20 mg of furosemide, intravenous bolus, followed by furosemide in endovenous continuous infusion, starting at 60 mg/day).
  The objective of this approach was to achieve negative fluid balance, between 600 to 1400 mL/day adjusted to body surface area, with a final target of 8-10% of body weight in up to 8 days. The furosemide dose was titrated considering heart rate and blood pressure, target fluid balance, hematocrit, and serum creatinine.
- NO-NEGBAL: Treatment for COVID-19 pneumonia in this series were based on standard recommendations.
  All patients in this group received dexamethasone 6 mg/day and thromboembolic prevention with enoxaparin 40 mg/day.
  Participants in the NO-NEGBAL group, did not received a NEGBAL approach as treatment.

SUMMARY:
In COVID-19, pulmonary edema has been attributed to "cytokine storm". However, it is known that SARS-CoV-2 promotes angiotensin-converting enzyme 2 deficiency, it increases angiotensin II and this triggers volume overload. The current study is based on patients with COVID-19, tomographic evidence of pulmonary edema and volume overload. These patients received a standard goal-guided diuretic (furosemide) treatment: Negative Fluid Balance (NEGBAL) approach. This retrospective observational study consists of comparing two groups. The cases show patients with COVID-19 and lung injury treated with NEGBAL approach comparing it to the control group consisting of patients with COVID-19 and lung injury receiving standard treatment. Medical records of 120 critically ill patients (60 in NEGBAL group and 60 in control group) were reviewed: demographic, clinical, laboratory, blood gas and chest tomography (CT) before and during NEGBAL.

Once NEGBAL strategy started, different aspects were evaluated: clinical, gasometric and biochemical evolution until the 8th day, tomography until the 12th day, ICU stay, hospital stay and morbidity and mortality until the 30th day.

DETAILED DESCRIPTION:
In December 2019, a new coronavirus, known as severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), emerged in Wuhan, China and spread throughout the world.

In COVID-19, pulmonary edema has been described; however, the dominant paradigm is focused on cytokine storm as responsible for lung injury and subsequent acute respiratory distress syndrome (ARDS). Not everyone agreed with this paradigm. Sinha et al. challenged the role of this cytokine storm given that median interleukin-6 (IL-6) levels in non-COVID patients ARDS were up to 200 times higher than in patients with severe COVID-19. Gattinoni et al. maintained that COVID-19 presented as an "atypical form" of ARDS. On the other hand, Kuba et al. and Imai et al. reported that angiotensin-converting enzyme 2 (ACE2) levels during a SARS-CoV infection are decreased. Furthermore, in patients with COVID-19, plasma levels of Angiotensin II are higher than in healthy population and stimulate an upregulation of aldosterone level, triggering sodium and water retention. SARS-CoV-2 enters through ACE2 and downregulates ACE2 expression so that this enzyme is unable to exert its protective effects. The dysregulated activity of the renin angiotensin aldosterone system (RAAS) is partly responsible for pulmonary edema in COVID-19. ACE2 is known for its effect as the main counter-regulatory mechanism for the renin-angiotensin aldosterone system (RAAS), which is an essential player in blood pressure control by retaining sodium and water and increasing the intravascular fluid volume. SARS-CoV-2 binds ACE2 and accelerates the degradation of ACE2, and thus decreases the counteraction of ACE2 on RAAS. The final effect is increasing reabsorption of sodium and water and subsequent volume overload. The RAAS can be envisioned as a dual function system in which the vasoconstrictor/proliferative or vasodilator/antiproliferative actions are primarily driven by the ACE-ACE2 balance. According to that, an increased ACE/ACE2 activity ratio generated by the downregulation action of SARS-CoV-2 on ACE2 will lead to increased Angiotensin II and increased catabolism of Angiotensin 1-7, towards vasoconstriction, endothelial dysfunction, prothrombosis, proinflammatory, and antinatriuretic effect.

Acute pulmonary edema is caused mostly by one of the following mechanisms: pulmonary venous pressure elevation-volume overload-or augmentation of the alveolar capillary membrane permeability-inflammation. In fact, both mechanisms sometimes coexist and the distinction is irrelevant. There are bibliographic references of pulmonary edema in COVID-19, as well as evidence of volume overload in COVID-19: Lang et al. describes frequent and pronounced vasculature in affected lung areas that may be suggestive of disordered vasoregulation. Eslami et al. observed increased cardiothoracic ratio and it is also described as right ventricular dilatation. In this setting, a different approach emerged: moderate or severe COVID-19 could experience a severe acute pulmonary edema with a "dual hit". A "first hit" of pneumonitis-augmentation of the alveolar capillary membrane permeability-can lead to low hydrostatic pressure pulmonary edema. The "second hit" is high pressure pulmonary edema, caused by increase of hydrostatic pressure secondary to volume overload, a result of dysregulation of the RAAS. This results in a "dual hit" that triggers severe acute pulmonary edema. If this edema is not solved, then a "third hit" appears with secondary inflammation, superinfection, fibrosis and finally the typical ARDS. Consequently, the study group looked for patients with pulmonary edema before ARDS was triggered. Cases of moderate and severe COVID-19 were searched, with tomographic evidence of pulmonary edema: dilated superior vena cava, large pulmonary arteries, diffuse interstitial infiltrates and dilated right ventricle. At the detection of pulmonary edema in patients with COVID-19, a standard treatment consisting of oral hydric restriction and diuretics (NEGBAL approach) was initiated. The effects of furosemide on pulmonary edema were well established decades ago. To date there is no evidence that had suggested the model of pulmonary edema and volume overload secondary to the dysregulation of the renin angiotensin aldosterone system in COVID-19. The objective of this study is to compare patients with COVID-19 undergoing NEGBAL approach with a control group of patients with COVID-19 of similar demographic, clinical, gasometric and tomographic characteristics. Medical records of 120 adult patients were reviewed: demographic; clinical, laboratory; Pro b-type natriuretic peptide (pro-BNP): (negative: below 125 pg/mL); high-sensitivity cardiac troponin (hs-cTnT): (negative: <14 ng/L); blood gas; chest tomography (CT); oxygen therapy support and mechanical ventilation (MV) requirements, all of which were reviewed and recorded by investigators. With the purpose of knowing the patient's basal hematocrit before COVID-19, prior hematocrit, if any, defined as hematocrit previous to COVID-19 infection (hematocrit prior to admission to NEGBAL) was also reviewed.

Once the NEGBAL strategy began, the clinical, tomographic, gasometric, biochemical evolution was evaluated until the 8th day (until the 12th day for tomography), ICU stay, hospital stay and morbidity and mortality until the 30th day.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patients subjected to NEGBAL group are as follows:

* confirmed diagnosis of COVID-19
* PaO2/FiO2 (ratio of arterial oxygen partial pressure to fractional inspired oxygen) <300;
* Patients over 18 years of age and
* tomographic evidence of acute pulmonary edema, defined as dilated superior vena cava, large pulmonary arteries, diffuse interstitial infiltrates with Kerley lines, and dilated right ventricle or dilated cardiac axis.

Patients subjected to NEGBAL underwent a treatment with furosemide in continuous intravenous infusion, guided by objectives: Negative Fluid Balance approach (NEGBAL).

Inclusion criteria for patients subjected to NO-NEGBAL-Control Group- are as follows:

* confirmed diagnosis of COVID-19 through real-time reverse transcriptase polymerase chain reaction (RT-PCR) assay with samples obtained from nasopharyngeal swab or positive antinucleocapsid immunoglobulin M (IgM) antibodies;
* ratio of arterial oxygen partial pressure to fractional inspired oxygen (PaO2/FiO2) <300;
* age older than 18 years, and
* tomographic evidence of acute pulmonary edema, defined as dilated superior vena cava, large pulmonary arteries, diffuse interstitial infiltrates with Kerley lines, and dilated right ventricle or dilated cardiac axis.

Patients subjected to NO-NEGBAL group, did not receive NEGBAL approach as treatment.

Exclusion Criteria for both groups are as follows:

* patients with prior indication of diuretics for another reason,
* renal failure,
* cardiac failure (diagnosis by echocardiography),
* hepatic failure,
* hypernatremia or hyponatremia,
* hypotension or shock.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population of patients with COVID-19 admitted to the ICU in a high complexity healthcare institution of Mar del Plata, Argentina.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-11-28 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Mortality | Until the 30th day after admission or discharge
  Mortality measured in days after admission
Oxygenation | From admission to day 7; until discharge, death, or until the 30th day, depending on which appears first.
  Evolution of oxygenation during hospitalization (measured by PaO2/FiO2). To analyze the correlation between the variation of the PaO2/FiO2 ratio and the NEGBAL variables, a linear regression model of the form PAFIBAL~β0+β1NEGBAL was used. For the model, the response variable PAFIBAL was registered as the difference in the PaO2/FiO2 between admission to NEGBAL to day 7. Continuous variables were expressed as means. Categorical variables were summarized as counts. No changes (adjustments) were made for missing data. The paired sample T test was used. All statistical tests were 2-tailed. A p-value < 0.05 was considered statistically significant. The analysis was not adjusted for multiple comparisons and given the possibility of a type I error, the findings should be interpreted as exploratory and descriptive. All analyses were performed using R software, version 4.1.1 (R Foundation for Statistical Computing)

SECONDARY OUTCOMES:
Number of participants with mechanical ventilation requirements (MV invasive) | Until discharge, death, or up to 30 days, depending on which appears first.
CT infiltrates | Prior to starting NEGBAL approach, between admission to day 4, day 8 and day 12 of NEGBAL.
  Evaluation of CT infiltrates, measured through the score described by Pan F et al, used as a semiquantitative measurement using the sum of lung involvement-5 lobes. Each lobe on a scale from 0 (normal) to 5 (maximum infiltrate) being the maximum CT score 25.
Measurement of the superior vena cava diameter | Prior to starting NEGBAL approach, between admission to day 4, day 8 and day 12 of NEGBAL.
  Measured in CT just above the arch of the azygos veins. Unit of measurement: millimeters (mm)
Measurement of cardiac axis diameter | Prior to starting NEGBAL approach, between admission to day 4, day 8 and day 12 of NEGBAL.
  Transverse measurement across the 4 cavities (in centimeters)

OTHER OUTCOMES:
Length of stay in ICU | Until discharge, death, or until the 30th day, depending on which appears first.
Length of hospital stay | Until discharge, death, or until the 30th day, depending on which appears first.

CONTACTS AND LOCATIONS:
Overall Officials: José LF Santos, MD, Principal Investigator — Clínica Colón - Mar del Plata - Argentina
Locations (1):
- Clínica Colón, Mar del Plata, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cui X, Chen W, Zhou H, Gong Y, Zhu B, Lv X, Guo H, Duan J, Zhou J, Marcon E, Ma H. Pulmonary Edema in COVID-19 Patients: Mechanisms and Treatment Potential. Front Pharmacol. 2021 Jun 7;12:664349. doi: 10.3389/fphar.2021.664349. eCollection 2021. PMID 34163357
- [Background] Xu Z, Shi L, Wang Y, Zhang J, Huang L, Zhang C, Liu S, Zhao P, Liu H, Zhu L, Tai Y, Bai C, Gao T, Song J, Xia P, Dong J, Zhao J, Wang FS. Pathological findings of COVID-19 associated with acute respiratory distress syndrome. Lancet Respir Med. 2020 Apr;8(4):420-422. doi: 10.1016/S2213-2600(20)30076-X. Epub 2020 Feb 18. No abstract available. PMID 32085846
- [Background] Rasch S, Schmidle P, Sancak S, Herner A, Huberle C, Schulz D, Mayr U, Schneider J, Spinner CD, Geisler F, Schmid RM, Lahmer T, Huber W. Increased extravascular lung water index (EVLWI) reflects rapid non-cardiogenic oedema and mortality in COVID-19 associated ARDS. Sci Rep. 2021 Jun 1;11(1):11524. doi: 10.1038/s41598-021-91043-3. PMID 34075155
- [Background] Kuebler WM, Jordt SE, Liedtke WB. Urgent reconsideration of lung edema as a preventable outcome in COVID-19: inhibition of TRPV4 represents a promising and feasible approach. Am J Physiol Lung Cell Mol Physiol. 2020 Jun 1;318(6):L1239-L1243. doi: 10.1152/ajplung.00161.2020. Epub 2020 May 13. PMID 32401673
- [Background] Sun X, Wang T, Cai D, Hu Z, Chen J, Liao H, Zhi L, Wei H, Zhang Z, Qiu Y, Wang J, Wang A. Cytokine storm intervention in the early stages of COVID-19 pneumonia. Cytokine Growth Factor Rev. 2020 Jun;53:38-42. doi: 10.1016/j.cytogfr.2020.04.002. Epub 2020 Apr 25. PMID 32360420
- [Background] Mangalmurti N, Hunter CA. Cytokine Storms: Understanding COVID-19. Immunity. 2020 Jul 14;53(1):19-25. doi: 10.1016/j.immuni.2020.06.017. Epub 2020 Jun 28. PMID 32610079
- [Background] Langer-Gould A, Smith JB, Gonzales EG, Castillo RD, Figueroa JG, Ramanathan A, Li BH, Gould MK. Early identification of COVID-19 cytokine storm and treatment with anakinra or tocilizumab. Int J Infect Dis. 2020 Oct;99:291-297. doi: 10.1016/j.ijid.2020.07.081. Epub 2020 Aug 6. PMID 32768693
- [Background] Hu B, Huang S, Yin L. The cytokine storm and COVID-19. J Med Virol. 2021 Jan;93(1):250-256. doi: 10.1002/jmv.26232. Epub 2020 Sep 30. PMID 32592501
- [Background] Fara A, Mitrev Z, Rosalia RA, Assas BM. Cytokine storm and COVID-19: a chronicle of pro-inflammatory cytokines. Open Biol. 2020 Sep;10(9):200160. doi: 10.1098/rsob.200160. Epub 2020 Sep 23. PMID 32961074
- [Background] Marini JJ, Gattinoni L. Management of COVID-19 Respiratory Distress. JAMA. 2020 Jun 9;323(22):2329-2330. doi: 10.1001/jama.2020.6825. No abstract available. PMID 32329799
- [Background] Sinha P, Matthay MA, Calfee CS. Is a "Cytokine Storm" Relevant to COVID-19? JAMA Intern Med. 2020 Sep 1;180(9):1152-1154. doi: 10.1001/jamainternmed.2020.3313. No abstract available. PMID 32602883
- [Background] Gattinoni L, Coppola S, Cressoni M, Busana M, Rossi S, Chiumello D. COVID-19 Does Not Lead to a "Typical" Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2020 May 15;201(10):1299-1300. doi: 10.1164/rccm.202003-0817LE. No abstract available. PMID 32228035
- [Background] Kuba K, Imai Y, Rao S, Gao H, Guo F, Guan B, Huan Y, Yang P, Zhang Y, Deng W, Bao L, Zhang B, Liu G, Wang Z, Chappell M, Liu Y, Zheng D, Leibbrandt A, Wada T, Slutsky AS, Liu D, Qin C, Jiang C, Penninger JM. A crucial role of angiotensin converting enzyme 2 (ACE2) in SARS coronavirus-induced lung injury. Nat Med. 2005 Aug;11(8):875-9. doi: 10.1038/nm1267. Epub 2005 Jul 10. PMID 16007097
- [Background] Imai Y, Kuba K, Rao S, Huan Y, Guo F, Guan B, Yang P, Sarao R, Wada T, Leong-Poi H, Crackower MA, Fukamizu A, Hui CC, Hein L, Uhlig S, Slutsky AS, Jiang C, Penninger JM. Angiotensin-converting enzyme 2 protects from severe acute lung failure. Nature. 2005 Jul 7;436(7047):112-6. doi: 10.1038/nature03712. PMID 16001071
- [Background] Liu Y, Yang Y, Zhang C, Huang F, Wang F, Yuan J, Wang Z, Li J, Li J, Feng C, Zhang Z, Wang L, Peng L, Chen L, Qin Y, Zhao D, Tan S, Yin L, Xu J, Zhou C, Jiang C, Liu L. Clinical and biochemical indexes from 2019-nCoV infected patients linked to viral loads and lung injury. Sci China Life Sci. 2020 Mar;63(3):364-374. doi: 10.1007/s11427-020-1643-8. Epub 2020 Feb 9. PMID 32048163
- [Background] Santos RA, Ferreira AJ, Simoes E Silva AC. Recent advances in the angiotensin-converting enzyme 2-angiotensin(1-7)-Mas axis. Exp Physiol. 2008 May;93(5):519-27. doi: 10.1113/expphysiol.2008.042002. Epub 2008 Feb 29. PMID 18310257
- [Background] Chen D, Li X, Song Q, Hu C, Su F, Dai J, Ye Y, Huang J, Zhang X. Assessment of Hypokalemia and Clinical Characteristics in Patients With Coronavirus Disease 2019 in Wenzhou, China. JAMA Netw Open. 2020 Jun 1;3(6):e2011122. doi: 10.1001/jamanetworkopen.2020.11122. PMID 32525548
- [Background] Connell JM, Davies E. The new biology of aldosterone. J Endocrinol. 2005 Jul;186(1):1-20. doi: 10.1677/joe.1.06017. PMID 16002531
- [Background] Vaduganathan M, Vardeny O, Michel T, McMurray JJV, Pfeffer MA, Solomon SD. Renin-Angiotensin-Aldosterone System Inhibitors in Patients with Covid-19. N Engl J Med. 2020 Apr 23;382(17):1653-1659. doi: 10.1056/NEJMsr2005760. Epub 2020 Mar 30. No abstract available. PMID 32227760
- [Background] Gurwitz D. Angiotensin receptor blockers as tentative SARS-CoV-2 therapeutics. Drug Dev Res. 2020 Aug;81(5):537-540. doi: 10.1002/ddr.21656. Epub 2020 Mar 4. PMID 32129518
- [Background] Ware LB, Matthay MA. Clinical practice. Acute pulmonary edema. N Engl J Med. 2005 Dec 29;353(26):2788-96. doi: 10.1056/NEJMcp052699. No abstract available. PMID 16382065
- [Background] Lang M, Som A, Carey D, Reid N, Mendoza DP, Flores EJ, Li MD, Shepard JO, Little BP. Pulmonary Vascular Manifestations of COVID-19 Pneumonia. Radiol Cardiothorac Imaging. 2020 Jun 18;2(3):e200277. doi: 10.1148/ryct.2020200277. eCollection 2020 Jun. PMID 34036264
- [Background] Eslami V, Abrishami A, Zarei E, Khalili N, Baharvand Z, Sanei-Taheri M. The Association of CT-measured Cardiac Indices with Lung Involvement and Clinical Outcome in Patients with COVID-19. Acad Radiol. 2021 Jan;28(1):8-17. doi: 10.1016/j.acra.2020.09.012. Epub 2020 Oct 1. PMID 33041195
- [Background] Argulian E, Sud K, Vogel B, Bohra C, Garg VP, Talebi S, Lerakis S, Narula J. Right Ventricular Dilation in Hospitalized Patients With COVID-19 Infection. JACC Cardiovasc Imaging. 2020 Nov;13(11):2459-2461. doi: 10.1016/j.jcmg.2020.05.010. Epub 2020 May 15. No abstract available. PMID 32426088
- [Background] Li YL, Zheng JB, Jin Y, Tang R, Li M, Xiu CH, Dai QQ, Zuo S, Wang HQ, Wang HL, Zhao MY, Ye M, Yu KJ. Acute right ventricular dysfunction in severe COVID-19 pneumonia. Rev Cardiovasc Med. 2020 Dec 30;21(4):635-641. doi: 10.31083/j.rcm.2020.04.159. PMID 33388009
- [Background] Patil VP, Salunke BG. Fluid Overload and Acute Kidney Injury. Indian J Crit Care Med. 2020 Apr;24(Suppl 3):S94-S97. doi: 10.5005/jp-journals-10071-23401. PMID 32704211
- [Background] Gluecker T, Capasso P, Schnyder P, Gudinchet F, Schaller MD, Revelly JP, Chiolero R, Vock P, Wicky S. Clinical and radiologic features of pulmonary edema. Radiographics. 1999 Nov-Dec;19(6):1507-31; discussion 1532-3. doi: 10.1148/radiographics.19.6.g99no211507. PMID 10555672
- [Background] Gandhi SK, Powers JC, Nomeir AM, Fowle K, Kitzman DW, Rankin KM, Little WC. The pathogenesis of acute pulmonary edema associated with hypertension. N Engl J Med. 2001 Jan 4;344(1):17-22. doi: 10.1056/NEJM200101043440103. PMID 11136955
- [Background] Pan F, Ye T, Sun P, Gui S, Liang B, Li L, Zheng D, Wang J, Hesketh RL, Yang L, Zheng C. Time Course of Lung Changes at Chest CT during Recovery from Coronavirus Disease 2019 (COVID-19). Radiology. 2020 Jun;295(3):715-721. doi: 10.1148/radiol.2020200370. Epub 2020 Feb 13. PMID 32053470
- [Background] Santos JLF, Zanardi P, Alo V, Rodriguez M, Magdaleno F, De Langhe V, Dos Santos V, Murialdo G, Villoldo A, Coria M, Quiros D, Milicchio C, Garcia Saiz E. Pulmonary Edema in COVID-19 Treated with Furosemide and Negative Fluid Balance (NEGBAL): A Different and Promising Approach. J Clin Med. 2021 Nov 28;10(23):5599. doi: 10.3390/jcm10235599. PMID 34884300